CLINICAL TRIAL: NCT03342833
Title: Blood Flow Restriction Training in Chronic Heart Failure: an Effective Training Strategy?
Acronym: BFR-CHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, KK Witte, Senior Lecturer in Cardiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17.YH.0348
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (Active Comparator)
  Interventions: Device: Blood flow restriction
- Usual training (Sham Comparator)
  Interventions: Device: Blood flow restriction

INTERVENTIONS:
Device: Blood flow restriction — Occlusion of venous flow between bouts of HIIT training exercise

SUMMARY:
The purpose of this current study proposal is to identify the potential physiological adaptations arising from a combined BFR+HIIT training intervention in CHF patients. We hypothesise that the addition of BFR to HIIT will increase whole-body V̇O2peak by promoting vascular and skeletal muscle adaptations above that seen with HIIT alone. The secondary outcomes of this study are to determine if such a training intervention leads to clinical improvements in exercise intolerance symptoms and quality of life indices. Given that the majority of previous research in to both BFR and HIIT has largely involved young, healthy and relatively active participants, the final objective of this current proposal is to determine the viability, tolerability and efficacy of these training modalities in an elderly cohort of predominantly sedentary CHF patients.

DETAILED DESCRIPTION:
Exercise training in CHF is a potentially effective intervention for improving symptomatic and prognostic outcomes, but remains underutilised in contemporary CHF management in the United Kingdom. This underutilisation may be partly the result of multiple approaches to training but also due to inconsistent and overall modest results of any of the interventions on important patient-orientated outcomes. A key consideration in this latter regard is whether disease related symptoms (e.g. dyspnoea) during exercise training limit the physiological work achievable during training, limiting the degree of the training stimulus to below the level at which physiological adaptation can be achieved. For example, in COPD participants only those in whom skeletal muscle fatigue was present after a training session evidenced any improvement in functional exercise capacity and health-related quality of life following a 3-month rehabilitation programme. Investigating novel approaches to training that promote greater gains in training effect may therefore lead to greater changes in patient-centred outcomes which will eventually stimulate greater uptake and alleviate the clinical burden chronic heart failure.

Blood Flow Restriction (BFR) training is a novel strategy in which a pressure cuff is inflated around the proximal portion of the exercising limbs (e.g. at the top of the arms or legs) during exercise or in recovery periods between exercise bouts. The pressure of the cuff is set to allow arterial blood flow but occlude venous return, subsequently altering (or maintaining) the local metabolic milieu, resulting in upregulation of several downstream pathways that augment the adaptive response to exercise. BFR has been successfully employed previously in combination with resistance exercise (RE) training to augment skeletal muscle hypertrophy in isolated peripheral muscles. Importantly, this training has been shown to promote muscle hypertrophy with concomitant increases in isokinetic strength in elderly individuals performing at low exercise work rates. This therefore demonstrates that BFR can induce comparatively similar adaptations at a lower power in elderly populations, suggesting this training strategy may have applications in other groups, such as CHF patients.

Additional studies have also demonstrated improvements in V̇O2peak by combining BFR with traditional low-intensity endurance training or high-intensity interval training (HIIT). Using a within-measures design, the first of these studies demonstrated that a 4-week training intervention (4 sessions per week) of 45-mins single-leg cycling under ischaemic conditions (induced by an external pressure of 50 mmHg in a pressure chamber) improved time-to-fatigue and V̇O2peak significantly more than an identical training intervention on the contralateral leg under normoxic (non-ischaemic) conditions. Further research with a between-measures design showed that 8-weeks of low-intensity cycling (40% V̇O2peak) with continuous BFR (160-210 mmHg) can increase both muscle strength and cross-sectional area as well as V̇O2peak significantly more than a control intervention using the same protocol without BFR. Interestingly, the control group exercised for longer during their training sessions (45-mins vs 15-mins for BFR) demonstrating that BFR not only has the potential to augment adaptations but is also a time-efficient modality of exercise. Given that lack of time is frequently cited as a barrier to regular exercise training, novel training interventions, such as BFR, that aren't time-consuming may be considered an attractive alternative form of exercise.

HIIT is also promoted as a time-efficient training modality that is known to promote comparable physiological adaptations to traditional high-volume low-intensity endurance exercise training. HIIT typically involves repeated bouts of intense ('near-maximal') exercise separated by brief periods of recovery. Some training studies have now combined BFR with HIIT (BFR+HIIT), applying the pressure cuff during recovery periods rather than during exercise. This combination of BFR+HIIT allows the working muscle to perform as normal during the short bouts of exercise; however, application of the cuff during recovery was shown to promote superior physiological adaptations above HIIT alone. Specifically, this study demonstrated that 4-weeks (2 sessions per week) of sprint interval training (4-7 bouts of maximal 30s cycling sprints with 4.5-mins recovery) combined with BFR (2-mins at 130 mmHg during the recovery period) significantly increased V̇O2peak compared to a control group performing the same training protocol without BFR.

Although the exact mechanisms responsible for this superior physiological response have yet to be fully elucidated, it is likely that the combination of BFR and HIIT promotes localized adaptations within the peripheral muscle tissues performing the exercise and then being subjected to BFR i.e. in the case of cycling, the quadriceps muscle group. Such adaptations are coordinated by the metabolic changes known to occur with both exercise and localized ischaemia. These result in an increased expression of several intracellular transcription factors, which subsequently orchestrate a cascade of downstream signalling pathways that promote physiological adaptations within skeletal muscle. These adaptations include increased capillarisation (angiogenesis), mitochondrial biogenesis, and a phenotypic switch towards predominantly slow-oxidative non-fatiguing type 1 muscle fibres. There has also been the suggestion that BFR can upregulate peripheral vascular adaptations. Collectively, these increase muscle oxygen delivery (̇Q̇mO2) and uptake (V̇mO2), both of which are now considered as crucial training-induced adaptive responses for increasing whole-body V̇O2peak and ameliorating exercise intolerance symptoms in CHF patients.

Indeed, several exercise training interventions in CHF patients have previously focused on promoting adaptive responses within the vasculature and peripheral skeletal muscles as a means of increasing V̇O2peak. The rationale for these studies is based on the poor correlation between LV ejection fraction and exercise intolerance symptoms in CHF. Furthermore, it is now well recognised that several peripheral impairments within the skeletal muscle system contribute to the symptoms of exercise intolerance in CHF. These include vascular dysfunction, muscle fibre atrophy, reduced capillarisation, mitochondrial dysfunction, and a shift towards predominantly fast-twitch glycolytic type IIx fibres. Collectively, these contribute to poor symptoms and therefore previous exercise training interventions in CHF patients have focused on promoting adaptations within the periphery as a means of increasing V̇O2peak and ameliorating exercise intolerance. Many of these studies have successfully demonstrated an increase in V̇O2peak primarily by promoting adaptations within the periphery. As such, we believe that BFR+HIIT represents a novel training stimulus that may promote adaptive responses within the vascular and skeletal muscle systems that are likely to have significant effects in terms of increasing V̇O2peak, ameliorating exercise intolerance and improving quality of life in CHF patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with New York Heart Association (NYHA) class II-III symptoms Stable CHF of at least 3 months duration On optimally tolerated medication for CHF No contraindications for cycling exercise Able and willing to give informed consent

Exclusion Criteria:

Class IV CHF Any contraindications to exercise Significant COPD (FEV1<60%), severe renal disease (eGFR<30), primary pulmonary hypertension as a co-morbidity Unable to give informed consent Current diagnosis of active cancer, inflammatory or musculoskeletal disease (e.g. rheumatoid arthritis), on-going infection or sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (ml.kg.min) | 4 weeks
  Peak oxygen consumption

SECONDARY OUTCOMES:
Quality of life (points) | 4 weeks
  Minnesota Living with Heart Failure Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR